CLINICAL TRIAL: NCT02160405
Title: Effect on Iron Levels by the Inclusion of Native Potato in the Diet of Children From 2 to 5 Years, ICBF Beneficiaries in the Municipalities of Carlosama, Cumbal, Guachucal, Túquerres y Pasto. Nariño. Colombia. Cluster Randomized Controlled Trial
Brief Title: Effect on Iron Levels by the Inclusion of Native Potato in the Diet of Children From 2 to 5 Years, ICBF Beneficiaries. Nariño. Colombia. Cluster Randomized Controlled Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidad Nacional de Colombia (Other)
Collaborators: McGill University (Other); Trade and Development Canada and Canadian International Development Agency (CIDA) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 74282013
Record Dates: First submitted 2014-05-08; First posted 2014-06-10 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-06

CONDITIONS: Effect on Iron Levels
Keywords: Iron levels

ARMS (1):
- Normal diet (Experimental)
  Interventions: Dietary Supplement: native potato

INTERVENTIONS:
Dietary Supplement: native potato

SUMMARY:
Nutritional deficiencies can lead to a number of health problems in children. In Latin America and the Caribbean countries, are registered so much problems of insufficient ingestion of food as of imbalances in the composition of the diet. These latter are expressed in the absence of micronutrients (iron, iodine, zinc, vitamin A), becoming a major health burden in developing countries. Being the globally's leading risk factor for disease and death, with hundreds of millions of pregnant women and young children particularly affected.

Justification: In Nariño, Colombia higher levels of malnutrition are presented with respect to country, just as micronutrient deficiency in children 1 to 4 years is higher than the national average. Most of these households are poor families with restrictions on access to food sources of these micronutrients, which is reported in a consumption of fruits, vegetables, milk products and meat, less than the national average. In this place is developing a project that aims to improve potato in higher yield, nutrition and resistance, for contribute to increase food security of native communities.

Objective: Evaluate the effect on iron levels generated by the inclusion of native potato in the diet of children aged 2-5 years in institutional beneficiaries modality ICBF, in the municipalities of Carlosama, Guachucal, Tuquerres, Cumbal and Pasto. Nariño. Colombia

Methods:

Design: A cluster randomized controlled trial. Open label Setting: 6 clusters, municipalities of Carlosama, Guachucal, Tuquerres, Cumbal and Pasto (two towns), which will be randomly assigned to 2 groups: the treatment group that receives native potato, and the control group that receives traditional potato, that will be include in the usual Institution meal Participants: children from 2 to 5 years, beneficiaries of programs in institutional modality of ICBF, in the municipalities of Carlosama, Guachucal, Tuquerres, Cumbal and Pasto.

Main outcome measures: serum ferritin and transferrin levels

The study was conducted in the form of institutional programs ICBF, in the municipalities of Carlosama, Guachucal, Túquerres, Cumbal and Pasto. Colombia. One hypothesis to a queue based on the changes that occur over time after surgery in the mean values (μ) of serum ferritin in the treatment group compared with the control group. A sample size of 212 children were calculated. The study has been presented and approved by the Ethics Committee of the Faculty of Medicine of the National University of Colombia and the Institutional Review Board of the participating institution. All parents of participating children must sign a written form to accept the voluntary participation of their child in the study.

DETAILED DESCRIPTION:
6 clusters, municipalities of Carlosama, Guachucal, Tuquerres, Cumbal and Pasto (two towns), which will be randomly assigned to 2 groups: the treatment group that receives native potato, and the control group that receives traditional potato, that will be include in the usual Institution meal

ELIGIBILITY:
Inclusion Criteria:

* children from 2 to 5 years, beneficiaries of programs in institutional modality of ICBF, in the municipalities of Carlosama, Guachucal, Tuquerres, Cumbal and Pasto

Exclusion Criteria:

* Children who met inclusion criteria but are not allowed to participate, refuse systematically to the test or don't go regularly to the institution

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 212 (Actual)
Dates: Start 2014-02; Primary Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
serum ferritin leves | 11 Weeks
Serum transferrin levels | 11 weeks

SECONDARY OUTCOMES:
Haemoglobin | 11 Weeks

OTHER OUTCOMES:
Weight | 11 weeks
Height | 11 Weeks
  Changes in Height over the time
food intake | 11 Weeks
  Changes in food intake in the period
supplement of micronutrient | 11 Weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Centros de Desarrollo Infantil Institucional, Pasto, Departamento de Nariño, Colombia